CLINICAL TRIAL: NCT02771041
Title: Prospective Randomized Assessment of the Influence of Early Preoperative Consultation on Satisfaction and the Average Length of Stay of Patients Who Underwent Total Hip Arthroplasty
Brief Title: Assessment of the Influence of Early Preoperative Consultation on Satisfaction and the Average Length of Stay of Patients Who Underwent Total Hip Arthroplasty
Acronym: PTHJ-8
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PTH J-8
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-05

CONDITIONS: Orthopedic Surgery
Keywords: Hip prothesis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group with D-8 medical consultation (Experimental): A medical consultation 8 days before surgery would serve to explain to the patient the early course of care, give advice and help to anticipate acts for its release "post-operative" as, for example, contact a physical therapist and a nurse or check to their community pharmacy if their heparin stock is enough and to answer any questions.
  Interventions: Procedure: medical consultation 8 days before surgery
- Group without D-8 medical consultation (No Intervention)

INTERVENTIONS:
Procedure: medical consultation 8 days before surgery — This consultation would serve to explain to the patient the early course of care, give advice and help to anticipate acts for its release "post-operative" as, for example, contact a physical therapist and a nurse or check to their community pharmacy if their heparin stock is enough and to answer any questions.
  Arms: Group with D-8 medical consultation

SUMMARY:
Arthroplastic hip surgery "fast-track" the subject of increasing interest and reduces the average length of stay and improve patient satisfaction. This fast circuit implemented in many schools uses dedicated inpatient units, preoperative patient education in multidisciplinary groups (including physiotherapists, nurses, rehabilitation doctors and surgeons), an analgesia protocol multimodal and a network dedicated to the outlet (1.2).

The investigators working hypothesis is that the mere realization of a preoperative visit a week before the intervention would reduce the average length of stay for all patients with a target of two nights (instead of 7.5 days currently) (3) to reduce the use of SSR during hospitalization. This consultation would serve to explain to the patient the early course of care, give advice and help to anticipate acts for its release "post-operative" as, for example, contact a physical therapist and a nurse or check to their community pharmacy if their heparin stock is enough and to answer any questions (Appendix 2: early information given to the patient consultation J-8).

The investigators protocol is inspired by the one already in place for outpatient PTH and PTH 1 night but invariably apply to all patients for whom a home is considered output.

DETAILED DESCRIPTION:
2. Objectives

1. Primary Objective Influence of preoperative consultation to "D-8" on the average length of stay of a randomized series multi-operator.
2. Secondary objectives

1. Evaluation of patient satisfaction and clinical status 2. Evaluation of the analgesic consumption 3. Evaluation of complications

3. Population concerned

1. Inclusion Criteria All patients undergoing total hip replacement
2. Exclusion criteria

1. Patient choosing immediately a supported SSR in postoperative 2. Geographical remoteness 3. Social isolation 4. Medical pathology requiring special monitoring (phlebitis history, coagulation disorders, anticoagulant therapy ...) 5. psychiatric pathology 6. Patients opting for the protocol "overnight"

4. Methodology and duration of the research This will be a prospective mono-centric multi-operator on the assessment of the management of patients in the surgical practice referred to above.

The inclusion of patients will take place over a period of 12 months, the goal is to include 90 patients (Figure 1).

Justification of Sample Size In 2013, for patients operated in a planned way, and with degenerative osteoarthritis, the length of stay was 7.5 days with a standard deviation of 3 days.

With such a length of stay, a staff of 2 to 45 subjects will detect a difference in length of stay of at least 1.8 days (significance level of 5%, 80% power). Such a difference is reasonably possible with the proposed organizational intervention.

Early preoperative consultation will be proposed to the randomized patient. When the patient is included in the group studied, it will be presented during the preoperative consultation early an information document with advice and guidance for patients to anticipate acts provided for its release "post-operative" (cf. . Appendix 2: patient information delivered early consultation J-8). This consultation will educate patients about what will happen when they leave, specifying concretely how their articulation with the city and the various professionals involved will have been planned and respond to all the issues raised.

Data collection Clinical data will be collected anonymously by an internal orthopedic surgery service for all patients included in the study by the realization of the Oxford hip score before the intervention (J-1), an assessment of pain through verbal validated scale (VAS), of St Joseph satisfaction questionnaire (validated questionnaire Saphora) accompanied by a verbal scale patient discharge and a telephone call 30 days after surgery to achieve again the Oxford hip score, evaluation of pain by VAS and patient satisfaction by simple verbal scale (see Annex 1) (4).

The criteria for hospital discharge are:

* Clinically: clean dressing, no fever, no comorbidity decompensation, EVA <4 with analgesics.
* Biologically: Hemoglobin> 10.
* Functionally: 3 steps climbing ability, ability to walk twenty meters and to go to the bathroom alone.

The assessment criteria will be used:

Primary endpoint:

- Average length of stay

Criterion of secondary judgments:

* Score Oxford Hip before and after the intervention
* Patient satisfaction (verbal scale: 0 to 10) before and after the intervention
* St. Joseph Satisfaction Questionnaire (validated questionnaire Saphora)
* Evaluation of pain by VAS before and after the intervention
* Morbidity and mortality

randomization: Randomization in the 2 groups (usual care without consultation with J-8 versus consultation with J-8) will be carried by the patient. The patient list will be balanced by randomly alternating blocks. orthopedic service personnel will not be notified in advance of schedule to avoid a bias in the management of patients with the service.

Data processing :

For each subject will be awarded an identifier (original name and surname - year of birth) and the data will be entered on a computer file which will be sent to the statistician in charge of analyzing the GHPSJ site. There will be no exchange of personal data.

Statistical analysis :

To find and test differences, univariate analyzes will use the test t-Student for continuous variables and the chi of 2 for categorical variables or their nonparametric equivalents. The significance level was set at p <0.05. If imbalance groups, a multivariate model is developed

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing total hip replacement

Exclusion Criteria:

1. Patient choosing immediately a supported SSR in postoperative
2. Geographical remoteness
3. Social isolation
4. Medical pathology requiring special monitoring (phlebitis history, coagulation disorders, anticoagulant therapy ...)
5. psychiatric pathology
6. Patients opting for the protocol "overnight"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Average length of stay | After surgery at Day 1

SECONDARY OUTCOMES:
OXFORD Score for Hip | Before and after surgery at Day -1 then Day 1
Patient satisfaction (verbal scale: 0 to 10) | Before and after surgery at Day -1 then Day 1
  Patient satisfaction (verbal scale: 0 to 10)
St. Joseph Satisfaction | After surgery when leaving the hospital, in average in the 3 Days
  St. Joseph Satisfaction Questionnaire (validated questionnaire Saphora)
Evaluation of pain by VAS | Before and after surgery at Day -1 then Day 1
  Evaluation of pain by VAS before and after the intervention
Morbidity | In the week after surgery
Mortality | In the week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume RIOUALLON, MD, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)